CLINICAL TRIAL: NCT04925635
Title: The Effect of Fistula Care Training With Mobile Health Application on Hemodialysis Patients' Adaptation and Self-Care Behaviors
Brief Title: Fistula Care and Mobile Health Applications in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Cevriye Ozdemir, Lecturer, Saglik Bilimleri Universitesi
Other Study IDs: i060708c.A
Record Dates: First submitted 2021-06-01; First posted 2021-06-14 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Nursing Caries; Arterio-venous Fistula; mHealth
Keywords: Hemodialysis; nursing; arteriovenous fistula; care; compliance; mobile health application
MeSH Terms: conditions — Arteriovenous Fistula; Patient Compliance | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: The arteriovenous fistula care mobile health application will be installed and promoted on the smart phones of the patients in the experimental group.
  Interventions: Behavioral: experimental group
- control group: Patients in the control group will receive arteriovenous fistula care training and a training booklet will be given.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: experimental group — The arteriovenous fistula care mobile health application will be installed and promoted on the smart phones of the patients in the experimental group. Arteriovenous fistula care mobile health application will be installed in daytime groups during working hours during or at the end of dialysis according to the patient's request. In addition, the information contained in the arteriovenous care mobile health application will be verbally explained to the patients and their relatives, as well as shown in practice. The training results were evaluated by the researcher in the 1st and 3rd months in the "Scale for Evaluation of Self-Care Behaviors Related to Arteriovenous Fistula in Hemodialysis Patients", "Final Level of Renal Failure Compliance Scale", "Arteriovenous Fistula Care Education Knowledge Level Evaluation Form (Post-Training Section)" and " Visual Benchmarking Scale ".
  Groups: experimental group
Behavioral: control group — Patients in the control group will receive arteriovenous fistula care training and a training booklet will be given. The information contained in the booklet will be explained orally to the patients and their relatives by the researcher, and will also be shown in practice. The results of the training were determined by the researcher at the 1st and 3rd months of the "Self-Care Behaviors Scale for Arteriovenous Fistula in Hemodialysis Patients", "End Stage Renal Failure Compliance Scale", "Arteriovenous Fistula Care Training Information Level Assessment Form (Post-training section)" and "Visual It will be evaluated with the "Comparison Scale".
  Groups: control group

SUMMARY:
In recent years, applications designed specifically to encourage physical activity in the field of mobile technology have gained momentum. As a result of the literature research, no examples of mobile health applications developed with educational content on fistula care, which hemodialysis-dependent patients can reach at any time and place, have not been found. Based on this, it was planned to increase the knowledge level of arteriovenous fistula care and examine their self-care behaviors and their adaptation to the disease with the mobile application developed with a focus on education on fistula care, which can be used independently by machine-dependent hemodialysis patients. In this context, it is aimed that dialysis patients will benefit especially in arteriovenous fistula care applications, thanks to the ever-increasing mobile applications in daily use with the developing technology. It is thought that the use of these technology-based trainings will be more comfortable, useful and encouraging for their own self-care. It is planned to be a guide for healthcare professionals.

DETAILED DESCRIPTION:
Chronic renal failure is a clinical picture characterized by chronic, progressive deterioration in metabolic and endocrine functions, in adjusting the fluid-electrolyte balance of the kidney as a result of a decrease in glomerular filtration value. When the glomerular filtration value decreases to 5-10 ml/minute, end-stage renal failure develops. Renal replacement therapies such as hemodialysis, peritoneal dialysis and kidney transplantation are applied in patients diagnosed with end-stage renal disease. Renal replacement therapies are life-sparing treatments and the most common method applied is hemodialysis. The success of dialysis, which is a highly effective medical technology, in saving lives is indisputable. Arteriovenous fistula opened for hemodialysis is the lifeline of sick individuals, and hemodialysis is a critical treatment method based on the vascular access pathway. In this context, compliance with treatment is of vital importance in individuals with a diagnosis of end-stage renal disease, and lack of vascular access can reduce its efficiency in a short time. Studies show that only 25% of hemodialysis patients can take care of themselves.

The inadequacy of the individual's knowledge and behaviors of arteriovenous fistula care impairs adherence to treatment, reduces the effectiveness of the treatment and increases the cost. Interventions that encourage changes in health behavior and encourage individuals to change their lifestyle should be integrated into daily life, and there should be support for when and where individuals can make decisions that may affect their health. Mobile technologies, such as smart mobile phones, that individuals regularly carry, can be an effective platform for encouraging health behavior change, especially since they are likely to be with the individual when they need it.

In recent years, applications designed specifically to encourage physical activity in the field of mobile technology have gained momentum. As a result of the literature research, no examples of mobile health applications developed with educational content on fistula care, which hemodialysis-dependent patients can reach at any time and place, have not been found. Based on this, it was planned to increase the knowledge level of arteriovenous fistula care and examine their self-care behaviors and their adaptation to the disease with the mobile application developed with a focus on education on fistula care, which can be used independently by machine-dependent hemodialysis patients. In this context, it is aimed that dialysis patients will benefit especially in arteriovenous fistula care applications, thanks to the ever-increasing mobile applications in daily use with the developing technology. It is thought that the use of these technology-based trainings will be more comfortable, useful and encouraging for their own self-care. It is planned to be a guide for healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Literate (can understand and speak Turkish),
* Do not have a diagnosed mental and psychological disease,
* Hearing or visually impaired,
* Open to communication and cooperation,
* Having arteriovenous fistula,
* Having a smart phone,
* Individuals willing to participate in the research will be included.

Exclusion Criteria:

* Those with arteriovenous graft,
* Those with a catheter,
* Those receiving peritoneal dialysis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of individuals with arteriovenous fistula who applied to Private Hope Dialysis Center and Private Almet Dialysis Center for hemodialysis between June 2020 and October 2020. In the study, the experimental and control groups were selected from two different dialysis centers in order to eliminate the bias and considering the control group's exposure to the interference.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
self-care behavior | 5 month
  Patients were informed about the Self-Care Behaviors Assessment Scale for Arteriovenous Fistula in Hemodialysis Patients. (The scale consisting of 16 items in total; Each item is scored according to the statements opposite. A minimum of 1 point indicates that the specified self-care behavior never develops, and the highest 5 points indicate that the specified self-care behavior always exists. The minimum score that can be obtained from the scale is 16, and the maximum score is 80.As the score increases, it is evaluated that the person's self-care behaviors are positive.)
adaptation to illness | 5 month
  Patients were informed about the End Stage Renal Failure Compliance Scale. (It consists of 5 chapters and 46 items. The total score that can be obtained from the scale varies between 0 and 1200. As the score obtained from the scale increases, the level of adherence to treatment increases.)
knowledge level | 5 month
  Patients were informed about the Arteriovenous Fistula Care Education Evaluation Form. (It states that there is no "0 point" information when scoring the form, but "1 point" information. The total score that can be obtained from the form varies between 0 and 13. The higher the score, the higher the AVF care knowledge level.)

CONTACTS AND LOCATIONS:
Overall Officials: Cevriye Ozdemir, Lecturer, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided